CLINICAL TRIAL: NCT03306953
Title: The Effect of Rectus Muscle Approximation at Cesarean Delivery on Postoperative Pain
Brief Title: The Effect of Rectus Muscle Approximation at Cesarean Delivery on Pain Perceived After Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Omran, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5678
Record Dates: First submitted 2017-10-06; First posted 2017-10-11 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rectus muscle approximation (Active Comparator): Three sutures will be done for the the purpose of rectus muscle approximation in cesarean section.
  Interventions: Procedure: Rectus muscle approximation
- Control (No Intervention): No approximation for the rectus muscle will be done for the control group in cesarean section.

INTERVENTIONS:
Procedure: Rectus muscle approximation — The surgeon will take sutures to approximate rectus muscles at the end of cesarean delivery.
  Arms: Rectus muscle approximation

SUMMARY:
This is a prospective randomized controlled study to determine the clinical outcome of rectus muscle re-approximation at Cesarean delivery.

DETAILED DESCRIPTION:
This is a prospective randomized controlled study to determine the clinical outcome of rectus muscle re-approximation at Cesarean delivery. Postoperative pain will be assessed in 2 groups. Rectus muscle approximation will be done to the first group. The second group will be the control group.

ELIGIBILITY:
Inclusion Criteria:

* Women who will undergo first elective cesarean section
* Singleton pregnancy

Exclusion Criteria:

* Previous abdominal or pelvic surgery
* Medical or psychiatric disease
* Previous pelvic inflammatory disease
* Obesity
* Allergy to analgesics

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Early pain score | 24 hours after cesarean section
  Early pain score will be assessed by an investigator for patients

SECONDARY OUTCOMES:
Late pain score | 48 hours after cesarean section
  Late pain score will be assessed by an investigator for patients

CONTACTS AND LOCATIONS:
Overall Officials: Eman F Omran, M.D., Principal Investigator — Cairo University
Locations (1):
- Department of Obstetrics and Gynecology, Kasr Al-Ainy hospital, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided